CLINICAL TRIAL: NCT06079957
Title: Additional Benefits of Neck Exercises in Addition to Ergonomic Training in Office Workers With Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/20
Record Dates: First submitted 2023-10-08; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Neck Pain
Keywords: neck pain, ergonomics, strengthening exercises, stretching, pain, burnout, range of motion, disability
MeSH Terms: conditions — Neck Pain; Pain; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Both groups will be recruited concurrently. both groups will recieve treatment
Who Masked: Outcomes Assessor
Masking Description: Single blind study; in which only analyst will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and ergonomic intervention group (Experimental): Patients will be explained about the procedure and informed consent will be taken.
  1. Individuals will be given a copy of ergonomic guidelines to follow which includes:
     * Organize workstation according to the primary , secondary and tertiary zones.
     * Place frequently used items within the reach of an arm.
     * Don't move head while reading documents instead raise or lower the eyes to read.
     * Correct the monitor height such that the top of the screen is at or slightly lower than eye level.
     * Keep reference material upright at desk.
     * Avoid slouched postural habits, sit upright.
     * Adjust chair height in such a way that it shouldn't compress the thigh.
     * Arm rest should be at elbow flexion of 90 degrees.
     * Phone must be cradled between neck and shoulder to avoid forward head posture.
  2. Neck exercises will be given
  Interventions: Procedure: Ergonomic training; Procedure: Neck Exercises
- Group B(Ergonomic intervention group) (Active Comparator): Patients will be explained about the procedure and informed consent will be taken.
  Individuals will be given a copy of ergonomic guidelines to follow which includes:
  * Organize workstation according to the primary , secondary and tertiary zones.
  * Place frequently used items within the reach of an arm.
  * Don't move head while reading documents instead raise or lower the eyes to read.
  * Correct the monitor height such that the top of the screen is at or slightly lower than eye level.
  * Keep reference material upright at desk.
  * Avoid slouched postural habits, sit upright.
  * Adjust chair height in such a way that it shouldn't compress the thigh.
  * Arm rest should be at elbow flexion of 90 degrees.
  * Phone must be cradled between neck and shoulder to avoid forward head posture.
  Interventions: Procedure: Ergonomic training

INTERVENTIONS:
Procedure: Ergonomic training — 1. Individuals will be given a copy of ergonomic guidelines to follow which includes:
  * Organize workstation according to the primary , secondary and tertiary zones.
  * Place frequently used items within the reach of an arm.
  * Don't move head while reading documents instead raise or lower the eyes to read.
  * Correct the monitor height such that the top of the screen is at or slightly lower than eye level.
  * Keep reference material upright at desk.
  * Avoid slouched postural habits, sit upright.
  * Adjust chair height in such a way that it shouldn't compress the thigh.
  * Arm rest should be at elbow flexion of 90 degrees.
  * Phone must be cradled between neck and shoulder to avoid forward head posture.
Procedure: Neck Exercises — Neck Exercises Strengthening exercises of Deep cervical flexors,rhomboids,lower Trapezius, Middle Trapezius, serratus anterior.
  Neck Stretching of Suboccipitals,Sternocleidomastoid ,Scalenes,Upper trapezius, Levator scapulae,Pectoralis major and minor.
  Arms: Exercise and ergonomic intervention group

SUMMARY:
Neck pain is a multifactorial disease and the factors related to neck pain are physical workloads, poor ergonomic work design and certain psychosocial factors. It arises due to disease of cervical spine and soft tissues of the neck, muscle spasm, falling asleep in awkward position, prolong working at computer desk with bent neck. The objective of the study is to compare the effects of neck exercises in addition to ergonomic training and ergonomic training alone on pain severity, neck disability, cervical range of motion and burnout in neck pain among office workers

DETAILED DESCRIPTION:
Neck pain remains the most common musculoskeletal disorder faced by office workers. There are an increasing number of reports available in regards to neck pain whether it is related with muscles, tendons, joints or soft tissue inflammation. It arises due to disease of cervical spine and soft tissues of the neck, muscle spasm, falling asleep in awkward position, prolong working at computer desk with bent neck. It has multiple treatment options and neck exercises are one of them. However, no concrete evidence is available on the effects of both neck exercises and ergonomic training on neck pain. this study will help individuals to maintain health and safety in the workplace while maintaining efficiency in their job performance by introducing proper ergonomic guidelines. This will eventually going to increase quality of work, productivity as a team and satisfaction with work. It will create awareness about utilization of ergonomic and exercise intervention without many side effects to avoid WMSDs. It will determine the emotional and psychological exhaustion among office workers with neck pain. It will supplement the existing literature. The main objectives of the study is to compare the effects of neck exercises in addition to ergonomic training and ergonomic training alone on pain severity, neck disability, cervical range of motion and burnout in neck pain among office workers.This RCT will be carried out in a period of one year (January 2023-2024). The sample size of 54 participants will be recruited according to inclusion and exclusion criteria. Both males and females aged between 25-50 years working for 7-9 hours with postural neck pain will be included in the study. the participants must have neck pain above 4 on NPRS and neck pain without radiculopathy. The ones fulfilling the criteria will be selected through non-probability purposive sampling and allocated in groups (A and B) through coin toss method. Group A will receive neck exercises along with ergonomic guidelines and group B will only follow the ergonomic guidelines. Participants of both groups will receive intervention for 3 weeks on alternate days. The data will be collected through numeric pain rating scale, neck disability index, cervical range of motion and Oldenburg burnout inventory. The data will be analyzed on SPSS 22.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female office workers.
* Age 25-50 years.
* Individuals with working hours duration of 7-9 hours.
* Individuals with postural neck pain.
* Individuals with neck pain above 4 on NPRS.
* Individuals with primary complaint of neck pain without radiculopathy.

Exclusion Criteria:

* History of trauma to neck.
* Bilateral upper limb symptoms.
* Prior surgery to cervical and upper thoracic spine.
* History of whiplash injury.
* Degenerative disc disease.
* Diminished or absent sensations to pinprick in upper limb dermatomes.
* Positive two or more neurological signs.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 3 weeks
  It is an 11 item self-rated scale. Participants rate their pain from 0 to 10. Score of 0 indicates no pain whereas 10 represents worst pain ever experienced. It has an excellent reliability with an ICC of 0.93-0.96.
Neck Disability Index Urdu version (NDI-U) | 3 weeks
  This is a 10 item questionnaire. This is a self-rated questionnaire to rate disability. Participants choose from an option from 0 to 5. Scoring is done by taking sum of all the answers. Score of 0 shows no disability whereas 50 indicate maximum level of disability. Score 0-4 indicates no disability, 5-14 indicates mild disability, 15-24 indicates moderate disability, 25-34 indicates severe disability and above 34 indicates that the person is completely disabled by the pain. It has an excellent reliability with an ICC of 0.88.
Cervical Range of Motion using Goniometer | 3 weeks
  A goniometer has 12-inch arms and a full circle body. It has one stationary arm and the second moving arm. Movement is performed and range of motion is measured. Goniometer will be used to measure flexion, extension, lateral flexion and rotation. It has an ICC of 0.83-0.98
Oldenburg Burnout Inventory (OLBI) | 3 weeks
  This is a 16 item questionnaire. It is also a self-rated questionnaire which is used to determine burnout level. Participants choose an option from 0 to 4 on a likert scale. Scores of question number 2,3,4,6,8,9,11,12 are reversed in order to find a true score. Scoring is done by taking a sum of all the answers. 0 indicates no burnout whereas score of 64 indicates highest level of burnout encountered by an individual.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan